CLINICAL TRIAL: NCT00881907
Title: Tissue Characterization in Teeth Treated With a Regeneration Protocol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Kenneth Hargreaves, Chair, Department of Endodontics, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20090152H
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Pulp Necrosis
Keywords: Regeneration (revascularization) of dental pulp; Immature Permanent Tooth With a Diagnosis of Pulpal Necrosis
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): Group A subjects will be asked to attend a recall visit 2 months following completion of the treatment visits.
  Interventions: Drug: Triple Antibiotic Paste
- Group B (Experimental): Group B subjects will be asked to attend a recall visit at 4 months following completion of the treatment visits.
  Interventions: Drug: Triple Antibiotic Paste
- Group C (Experimental): Group C subjects will be asked to attend a recall visit at 6 months following completion of the treatment visits.
  Interventions: Drug: Triple Antibiotic Paste

INTERVENTIONS:
Drug: Triple Antibiotic Paste — ciprofloxacin, metronidazole & minocycline mixed to a 1:1:1 powder used as a intracanal medicament for disinfection and cell proliferation.
  Arms: Group A
Drug: Triple Antibiotic Paste — ciprofloxacin, metronidazole & minocycline mixed to a 1:1:1 powder used as a intracanal medicament for disinfection and cell proliferation.
  Arms: Group B
Drug: Triple Antibiotic Paste — ciprofloxacin, metronidazole & minocycline mixed to a 1:1:1 powder used as a intracanal medicament for disinfection and cell proliferation.
  Arms: Group C

SUMMARY:
The purpose of the investigators study is to characterize the composition of the hard and soft tissues present in root canals of teeth previously diagnosed with necrotic pulps and incomplete root formation and treated with a triple antibiotic regeneration protocol. The investigators hypothesis is that treatment of teeth with necrotic pulps and immature apices with triple antibiotic paste will stimulate continued root formation by the deposition of dentin at the root apices. The primary outcome measure will be histological identification of mineralized tissue and adherent cells in the apical third of these teeth.

DETAILED DESCRIPTION:
'Regeneration' as referred to in this protocol refers to the stimulation of continued root formation by the deposition of apical tissues subsequent to disinfection of a necrotic root canal and its contents and creation of a scaffold upon which cells can proliferate. While the proposed treatment protocol is currently being used in clinical practice and has been shown to be successful in case reports and case series, the nature of the proliferating apical tissues remains unknown. Thus, this study is uniquely positioned to address a critical gap in knowledge in the regeneration of a functional pulp-dentin complex. Moreover, results obtained from pediatric cases may well provide the essential foundation of knowledge for endodontists to apply this knowledge to the more difficult situation of regenerating the pulp-dentin complex of the full mature permanent tooth.

ELIGIBILITY:
Inclusion Criteria:

* Patient Inclusion Criteria:

  * Healthy volunteers ages 10-60 with a non-restorable (as determined by referring dentist), permanent tooth with a necrotic pulp and incomplete root development.
  * Persons who seem to be cooperative with dental treatment and able to indicate willingness to obtain treatment and participate in the study and who are capable of verbally expressing dissent.
  * Parents who express understanding of study treatments and consent to treatment for their child of the regenerative procedure.
  * Healthy patients (ASA Class I or II physical status) with no systemic health problems that may interfere with healing and cell growth.
* Tooth inclusion criteria:

  * Permanent tooth with necrotic pulp and immature root development, scheduled for extraction due to non-restorability.
  * Clinically confirmed necrotic pulp that will be confirmed with common endodontic pulp vitality tests (No response to cold or electric pulp test).
  * Clinically confirmed immature root development that will be assessed radiographically to confirm the non-restorability as diagnosed by the referring dentist.

Exclusion Criteria:

* Patient Exclusion Criteria:

  * Parents and patients unable to give consent or express dissent.
  * Patients who are unwilling to undergo the dental treatment.
  * Patients affected by temporomandibular joint disorders.
  * Patients affected by known orofacial pain disorders.
  * Patients with ASA Class III or IV physical status (Immuno-compromised patients including patients who self-report that they are an HIV carrier, undergoing steroid therapy or chemotherapy, or those who self-report with genetic or systemic diseases that could result in reduced immune response).
* Tooth Exclusion Criteria:

  * Teeth with vertical cracks that extend below the cemento-enamel junction.
  * Teeth that cannot be isolated using a rubber dam.
  * Teeth with non-odontogenic pathology.
  * Teeth whose apices are fully developed, as determined radiographically and correlated with dental age of patient.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be histological identification of mineralized tissue and adherent cells in the apical third of these teeth. | three year

SECONDARY OUTCOMES:
The secondary outcome measure will be conducted by measuring markers of stem cells prior to and after the formation of the blood clot. | three year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Hargreaves, DDS,PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States